CLINICAL TRIAL: NCT02722824
Title: Efficacy Investigation of a Non-invasive Wearable Electrostimulation Device for Alleviation of Parkinson's Disease Symptoms
Brief Title: Efficacy of a Non-invasive Device for Alleviation of Parkinson's Disease Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasemin Gürsoy Özdemir, Professor, Koç University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Par-01
Record Dates: First submitted 2016-03-06; First posted 2016-03-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Parkinson's Disease
Keywords: motor symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Wearable stimulators will be placed on the patients and controls without stimulation for 20 minutes
  Interventions: Other: Placebo
- Active Stimulation (Experimental): Instrinsic auricular muscles will be stimulated for 20 minutes
  Interventions: Device: Electro-stimulation
- Sham (Sham Comparator): An area out of the instrinsic auricular muscles region will be stimulated with the same parameters of the active group for 20 minutes
  Interventions: Device: Electro-stimulation
- Passive Control (No Intervention): Only the electrodes of the wearable stimulators will be inserted but there will not be electrostimulation for 20 minutes

INTERVENTIONS:
Device: Electro-stimulation
  Arms: Active Stimulation; Sham
Other: Placebo
  Arms: Placebo

SUMMARY:
Investigation efficacy of a non-invasive wearable electrostimulator device where the supplementary motor area, premotor area and/or subthalamic nucleus are stimulated bilaterally and extracranially.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* H&Y Stage >= 2
* Existing bradykinesia symptoms
* Existence of one of the symptoms below
* Resting Tremor
* Rigidity
* Walking disorder

Exclusion Criteria:

* Cardiac Pacemaker
* Psychiatric diagnosis
* Irregular heart/respiration rate
* Pregnancy
* Alcohol consumption
* Cardiovascular disease history
* Wearing an electro-active prosthesis
* Brain surgery history
* Ongoing TENS/PENS therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in the UPDRS Motor Score (Part III) | 10 minutes after the stimulation is initiated.
  Evaluation of patients' disease level with UPDRS examination at the middle of the stimulation
Change in the UPDRS Motor Score (Part III) | 30 minutes after the stimulation is terminated.
  Evaluation of patients' disease level with UPDRS examination 30 minutes after the stimulation is terminated.

SECONDARY OUTCOMES:
Change in the gait and balance parameters (cadence) | 10 minutes after the stimulation is initiated.
  cadence
Change in the gait and balance parameters (Stride length) | 10 minutes after the stimulation is initiated.
  Stride length in meters
Change in the gait and balance parameters (Stride velocity) | 10 minutes after the stimulation is initiated.
  Stride velocity in m/s
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Arm Swing Rate
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Arm Range of Motion
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Sit to Stand Duration
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Sit to Stand Peak Trunk Velocity
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Sit to Stand Peak Trunk Angle
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Leg Swing Rate
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Leg Range of Motion
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Turn to Sit Peak Turn Velocity
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Turn-to-Sit Trunk Range of Motion in Sagittal Plane
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Knee Range of Motion
Change in the gait and balance parameters | 10 minutes after the stimulation is initiated.
  Trunk Joint Angles
Change in the gait and balance parameters (cadence) | 30 minutes after the stimulation is terminated.
  cadence
Change in the gait and balance parameters (Stride length) | 30 minutes after the stimulation is terminated.
  Stride length in meters
Change in the gait and balance parameters (Stride velocity) | 30 minutes after the stimulation is terminated.
  Stride velocity in m/s
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Arm Swing Rate
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Arm Range of Motion
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Sit to Stand Duration
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Sit to Stand Peak Trunk Velocity
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Sit to Stand Peak Trunk Angle
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Leg Swing Rate
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Leg Range of Motion
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Turn-to-Sit Peak Turn Velocity
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Turn-to-Sit Trunk Range of Motion
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Knee Range of Motion
Change in the gait and balance parameters | 30 minutes after the stimulation is terminated.
  Trunk Joint Angles

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul
  - Koc University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided